CLINICAL TRIAL: NCT00606554
Title: A Randomized Controlled Trial of Computer-Driven Weaning Compared With Standard of Care Weaning in Medical Patients Requiring Mechanical Ventilation
Brief Title: Clinical Trial of a Computer-driven Weaning System for Patients Requiring Mechanical Ventilation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment of subjects
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-26906
Record Dates: First submitted 2008-01-03; First posted 2008-02-04 (Estimated); Results first posted 2011-08-17 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-11

CONDITIONS: Respiratory Insufficiency
Keywords: Respiratory Insufficiency; Ventilators, Mechanical; Ventilator Weaning; Therapy, Computer-Assisted
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Computer-assisted weaning (Experimental): Group assigned to the computer-assisted weaning program
  Interventions: Device: Computer-assisted weaning program
- Standard of care weaning (Active Comparator): Group assigned to receive current, evidence-based, standard of care for discontinuation of mechanical ventilation.
  Interventions: Behavioral: Standard of Care weaning

INTERVENTIONS:
Device: Computer-assisted weaning program — Closed-loop, knowledge-based, computer-assisted wean program initiated at the start of ventilator weaning.
  Other Names: Drager Evita Smartcare System
  Arms: Computer-assisted weaning
Behavioral: Standard of Care weaning — Evidence-based standard of care weaning process.
  Arms: Standard of care weaning

SUMMARY:
The purpose of this study is to compare the efficacy of a computer-assisted ventilator weaning system (Drager Smartcare) to our current standard of care in the medical intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Initiated on mechanical ventilation via endotracheal tube
* Admitted to Medical Intensive Care Unit and Medical Intensive Care Unit Team (Harrison Avenue Campus, Menino Pavilion)
* Requiring mechanical ventilation for more than 48 hours
* Meets prespecified weaning criteria

Exclusion Criteria:

* Do Not Resuscitate/Do Not Intubate order
* Pregnancy
* Mechanical ventilation initiated at another hospital
* Cardiac arrest for more than 5 minutes with poor neurologic prognosis
* Tracheostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine C Reardon, MD, Principal Investigator — Boston University
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

REFERENCES:
- See also: BUMC Pulmonary Center Home Page — http://www.bumc.bu.edu/pulmonary

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment start 1/2008 recruitment end: 5/2010 Recruited from Medical Intensive Care Unites Boston medical Center
Groups:
- Computer-assisted Wean: Group assigned to the computer-assisted weaning program Intervention Group
- Standard of Care: Group assigned to receive current, evidence-based, standard of care for discontinuation of mechanical ventilation.
  Comparator group
Period: Overall Study
Arm/Group | Computer-assisted Wean | Standard of Care
Started | 15 | 18
Completed | 15 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Computer-assisted Wean | Standard of Care | Total
Number analyzed (Participants) | 15 | 18 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (21) | 60.5 (15.5) | 55.7 (18.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 10 | 11 | 21
APACHE II Score [Mean (Standard Deviation); unit: score] — Acute Physiology and Chronic Health Evaluation Score Range 0-72 Higher score indicates more severe illness
  score | 23.3 (7.7) | 26.5 (7.1) | 25 (7.4)

OUTCOME MEASURES:

1. Primary Outcome: Duration of Weaning
Description: Duration of weaning was assessed as the time from the initiation of weaning (randomization) to the time of successful extubation (defined as 48 hours free of mechanical ventilation). Patients were followed for the duration of hospitalization and the time of weaning onset and successful liberation from the ventilator was noted.
Time Frame: Continuous (median weaning duration was 2 days)
Population: ITT
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Computer-assisted Wean | Standard of Care
Number analyzed (Participants) | 15 | 18
Days | 1.92 [0.98 to 4.78] | 2.15 [0.92 to 9.10]
Statistical Analysis 1: Comparison: Computer-assisted Wean vs Standard of Care; Test type: Superiority or Other; p = 0.60, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Duration of ICU Stay
Description: Duration of ICU stay after weaning initiation
Time Frame: from start of weaning to discharge from ICU, on average 1-2 weeks
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Computer-assisted Weaning | Standard of Care Weaning
Number analyzed (Participants) | 15 | 18
days | 10.2 [7.6 to 19.7] | 15 [7.9 to 20.3]

3. Secondary Outcome: Duration of Mechanical Ventilation
Description: Duration of mechanical ventilation from weaning initiation
Time Frame: from start of weaning to liberation from ventilator, on average 1-2 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Computer-assisted Wean | Standard of Care
Number analyzed (Participants) | 15 | 18
days | 1.91 [0.98 to 4.78] | 2.15 [0.92 to 9.1]

4. Secondary Outcome: Duration of Hospitalization
Time Frame: from start of weaning to discharge from hospital, on average 1-2 weeks
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Computer-assisted Wean | Standard of Care
Number analyzed (Participants) | 15 | 18
days | 19.1 [11.1 to 27.8] | 19.7 [15.7 to 25.4]

5. Secondary Outcome: Inpatient Mortality
Description: proportion of patients in each arm who died in the hospital
Time Frame: 28 days
Population: ITT
Measure: Number; unit: Participants
Groups:
- Computer-assisted Weaning: Group assigned to the computer-assisted weaning program. Intervention Group
- Standard of Care Weaning: Group assigned to receive current, evidence-based, standard of care for discontinuation of mechanical ventilation. Comparator group
Arm/Group | Computer-assisted Weaning | Standard of Care Weaning
Number analyzed (Participants) | 15 | 18
Participants | 1 | 6
Statistical Analysis 1: Comparison: Computer-assisted Weaning vs Standard of Care Weaning; Test type: Superiority or Other; p = 0.06, Chi-squared

6. Secondary Outcome: Sedation Requirements
Description: measure was not recorded
Time Frame: during weaning, on average 1-2 days
Population: Data were not recorded
Arm/Group | Computer-assisted Wean | Standard of Care
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Spontaneous Breathing Trials Prior to Extubation
Time Frame: from start of weaning to liberation from ventilator, on average 1-2 days
Measure: Median (Inter-Quartile Range); unit: SBTs
Arm/Group | Computer-assisted Wean | Standard of Care
Number analyzed (Participants) | 15 | 18
SBTs | 0 [0 to 1] | 1 [0 to 1]

8. Secondary Outcome: Complications (Death During Wean, Ventilator-associated Pneumonia During Wean, Self Extubation, Re-intubation)
Description: This outcome is a composite outcome of the total number of participants with any one of the above-listed weaning-associated complications.
Time Frame: Duration of weaning (median 2 days)
Population: Number of participants with adverse event during weaning
Measure: Number; unit: Participants
Arm/Group | Computer-assisted Wean | Standard of Care
Number analyzed (Participants) | 15 | 18
Participants | 7 | 8
Statistical Analysis 1: Comparison: Computer-assisted Wean vs Standard of Care; Test type: Superiority or Other; p = 0.90, Chi-squared

ADVERSE EVENTS:
Time Frame: Duration of hospitalization after initiation of mechanical ventilation. Median 20 days
Arm/Group | Computer-assisted Wean | Standard of Care
All-Cause Mortality (participants affected / at risk) | 1/15 | 6/18
Serious Adverse Events (participants affected / at risk) | 7/15 | 8/18
Other Adverse Events (participants affected / at risk) | 1/15 | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Computer-assisted Wean (N=15) | Standard of Care (N=18)
Need for Tracheostomy (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) — unable to be weaned from ventilator, required tracheostomy for long term ventilation
Ventilator associated pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Death during weaning process (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Re-intubation (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4) — required placement back on mechanical ventilator using endotracheal tube after intial extubations
Self-extubation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — patient removed endotracheal tube prior to physician order.
Non-invasive ventilation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) — received non-invasive mechanical ventilator through a mask after extubation
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Computer-assisted Wean (N=15) | Standard of Care (N=18)
High pressure support level reached (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — In one participant with a baseline PaCO2 level > 60mmHg, the computer-driven weaning system (SmartCare) increased delivered pressure support to 40cm H2O in an attempt to decrease end tidal CO2 to less then 60. No adverse clinical outcomes resulted.

LIMITATIONS AND CAVEATS:
This trial was terminated early due to slow recruitment. It did not reach the target N of 220.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No